CLINICAL TRIAL: NCT01869322
Title: Acute Management of Humeral Shaft Fractures: Sling vs. Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Darin Friess, M.D., M.P.H., Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009456
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Fracture of Shaft of Humerus
Keywords: Humerus; Fracture; Sling; Splint; Coaptation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling and Swathe (Experimental): In this arm, study subjects will receive sling and swathe immobilization for humeral shaft fracture.
  Interventions: Device: Sling and Swathe
- Coaptation Splint (Active Comparator): In this arm participants receive a coaptation splint for humeral shaft fracture.
  Interventions: Device: Coaptation Splint

INTERVENTIONS:
Device: Sling and Swathe — Sling and Swathe immobilization of humeral shaft fracture.
  Arms: Sling and Swathe
Device: Coaptation Splint — Coaptation splint immobilization of humeral shaft fractures.
  Arms: Coaptation Splint

SUMMARY:
When people break their arm and arrive at Oregon Health and Science University's Emergency Department (OHSU ED), they are treated with a short-term means of immobilizing their broken arm. The two most common ways of stabilizing the broken parts of the arm are 1) with a plaster-based coaptation splint, or 2) with a soft cloth sling and swathe. These hold the arm steady until the patient can schedule an appointment with the OHSU Orthopaedic Trauma clinic where they will receive definitive evaluation and stabilization/fixation. In much of the orthopaedic literature coaptation splints are the default immobilization method. The investigators hypothesize however, that sling and swathe immobilization may be equally effective for short term stabilization, while being faster to apply, and more comfortable for the patient. This randomized, unblinded prospective study will follow the satisfaction, quality of life and limited functional outcomes of all enrolled participants during the first week following their injury.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* acute midshaft humeral fracture within 48 hours

Exclusion Criteria:

* ED presentation more than 48 hours after injury
* Head injury
* Open fracture
* Pathological fracture
* Known pregnancy
* Inmate or prisoner
* Non-English speaking
* Sexual Assault (SA) victim
* Patient and Legally Authorized Representative unable to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 5 days
  Satisfaction questionaires will be administered 5 days after admission/enrollment in the study, or before any surgical fixation which occurs more than 48 hours after admission.

SECONDARY OUTCOMES:
Patient Pain | 5 days
  Patient narcotic usage and NRS pain score will be collected 5 days from admission/enrollment, or before any surgical fixation which occurs more than 48 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Darin Friess, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States